CLINICAL TRIAL: NCT04250194
Title: Navigation Endoscopy to Reach Indeterminate Lung Nodules Versus Trans-Thoracic Needle Aspiration, a Randomized Controlled Study (VERITAS)
Brief Title: Navigation Endoscopy to Reach Indeterminate Lung Nodules Versus Trans-Thoracic Needle Aspiration
Acronym: VERITAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Fabien Maldonado, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC THO 19102; NCI-2020-00632 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Lung Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Navigation Bronchoscopy (NB) with F-Nav (Experimental)
  Interventions: Device: Navigation bronchoscopy
- CT-guided Biopsy (Experimental)
  Interventions: Device: CT-Guided Biopsy

INTERVENTIONS:
Device: CT-Guided Biopsy — Images will be generated by a CT scanner to accurately insert a needle into the lung nodule allowing a sample to be removed for testing
  Arms: CT-guided Biopsy
Device: Navigation bronchoscopy — A virtual three-dimensional map of the lung will be generated enabling the physician to perform an anatomically precise biopsy
  Arms: Navigation Bronchoscopy (NB) with F-Nav

SUMMARY:
This study will evaluate which procedure is the best for patients referred for biopsy of a lung nodule (growth in the lung) meeting the size and location requirements of the protocol. Two different procedures are available for lung nodule biopsy:

1. a computed tomography guided biopsy ("CT-guided biopsy") which consists of sampling the nodule from the "outside-in", through the chest wall with CT guidance, and
2. navigation bronchoscopy, which is a procedure using technology designed to guide a catheter through the natural airway route (wind-pipe and bronchi) to access the nodule.

DETAILED DESCRIPTION:
Endpoints:

Primary:

• To evaluate diagnostic accuracy through 12 months of clinical follow-up

Secondary:

* To evaluate rate of pneumothorax.
* To evaluate rate of pneumothorax requiring chest tube placement.
* To evaluate clinically significant bleeding (defined by bleeding requiring intervention).
* To evaluate need for hospitalization after procedure.
* To evaluate duration of the procedure.
* To evaluate procedural factors associated with improved yield (type of biopsy, number of biopsies, use of radial ultrasound, presence of a bronchus sign, biopsy site).
* To evaluate need for additional nodule biopsy.
* To evaluate need for additional procedure for staging.
* To evaluate radiation exposure from fluoroscopy-guided bronchoscopy and CT for CT-guided biopsy.
* To evaluate need for F-Nav (digital tomosynthesis) during navigation bronchoscopy.
* To evaluate diagnostic yield
* To evaluate the rate at which the biopsy procedure yields a confident clinical diagnosis (including any added yield from endobronchial ultrasound-guided mediastinal and/or hilar lymph node biopsies or microbiologic studies which yield an explanation for a nodule despite non-diagnostic biopsy specimens).

ELIGIBILITY:
Inclusion Criteria:

* Patient is referred for biopsy of a single indeterminate pulmonary nodule, with the following characteristics regarding size, location, accessibility, and probability of malignancy:

  * Intermediate pre-test probability of malignancy as defined by a pre-test probability of malignancy between 10% and 100%, using a validated clinical prediction model, which is either:

    * The Brock model14 if no PET scan data are available, or
    * The Herder model15 if PET-CT data are available.
  * Size between 10 and 30 mm (long diameter).
  * Location peripheral, here defined as occupying the middle or outer third lung zones.
  * Accessible via navigation bronchoscopy and also accessible via CT-guided biopsy (i.e. the nodule is clinically suited to equal access by either procedure), as confirmed by an independent interventional panel.

Exclusion Criteria:

* Patients with proximal nodules, as defined by nodules present in the proximal 1/3 of the lung by dedicated software analysis (described below) will not be eligible for the study.
* Patients with multiple nodules requiring biopsy (patients may have other nodules not considered for biopsy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (7):
- United States (7):
  - University of California, San Diego, San Diego, California
  - Kootenai Health, Coeur d'Alene, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Lentz RJ, Frederick-Dyer K, Planz VB, Koyama T, Aboudara MC, Avasarala SK, Casey JD, Cheng GZ, D'Haese PF, Duke JD, Grogan EL, Hoopman TC, Johnson J, Katsis JM, Kurman JS, Low SW, Mahmood K, Rickman OB, Roller L, Salmon C, Shojaee S, Swanner B, Wahidi MM, Walston C, Silvestri GA, Yarmus L, Rahman NM, Maldonado F; Interventional Pulmonary Outcomes Group. Navigational Bronchoscopy or Transthoracic Needle Biopsy for Lung Nodules. N Engl J Med. 2025 Jun 5;392(21):2100-2112. doi: 10.1056/NEJMoa2414059. Epub 2025 May 18. PMID 40387025
- [Derived] Lentz RJ, Frederick-Dyer K, Planz VB, Koyama T, Aboudara MC, Swanner B, Roller L, Low SW, Salmon C, Avasarala SK, Hoopman TC, Wahidi MM, Mahmood K, Cheng GZ, Katsis JM, Kurman JS, D'Haese PF, Johnson J, Grogan EL, Walston C, Yarmus L, Silvestri GA, Rickman OB, Rahman NM, Maldonado F. Navigational Bronchoscopy versus Computed Tomography-guided Transthoracic Needle Biopsy for the Diagnosis of Indeterminate Lung Nodules: protocol and rationale for the VERITAS multicenter randomized trial. medRxiv [Preprint]. 2023 Nov 23:2023.11.22.23298915. doi: 10.1101/2023.11.22.23298915. PMID 38045245

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 288 participants were consented, 30 participants were excluded prior to randomization:
  * Failed central adjudication of procedure feasibility (n=20)
  * Withdrawal of informed consent (n=5)
  * New data available meeting exclusion criterion (n=5)
Period: Overall Study
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Started | 129 | 129
Completed | 121 | 113
Not Completed | 8 | 16
Not completed — Declined to schedule biopsy | 6 | 10
Not completed — Medically Unfit for Biopsy | 2 | 1
Not completed — New data available meeting exclusion criterion: PET/CT with avid adenopathy | 0 | 2
Not completed — New data available meeting exclusion criterion: interim CT demonstrated rapid growth to >30 mm | 0 | 2
Not completed — New data available meeting exclusion criterion: PET/CT with avid endobronchial lesion | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy | Total
Number analyzed (Participants) | 121 | 113 | 234
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [62 to 72] | 68 [61 to 74] | 67 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 64 | 57 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 121 | 110 | 231
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 110 | 105 | 215
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Comorbidities [Count of Participants; unit: Participants]
  Current or prior malignancy | 46 | 55 | 101
  Chronic Obstructive Pulmonary Disease (COPD) | 49 | 48 | 97
  Coronary artery disease | 25 | 16 | 41
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.6 [23.9 to 31.5] | 27.9 [24.0 to 31.2] | 27.7 [24.0 to 31.3]
Tobacco smoking history [Count of Participants; unit: Participants]
  Current | 39 | 24 | 63
  Former | 55 | 66 | 121
  Non-smoker | 27 | 23 | 50
Pack-years [Median (Inter-Quartile Range); unit: pack-years] | 43 [20 to 55] | 35 [20 to 47] | 40.0 [20.0 to 52.0]

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Proportion of biopsies leading to a definitive diagnosis, comparing the bronchoscopy pathway to the CT-guided biopsy pathway. Definitive diagnoses are pre-defined as any of the following:
  * Malignant, OR
  * Abnormal tissue (excluding normal or absence of lung parenchyma) followed by a surgical lung biopsy yielding the same histological diagnosis, OR
  * Specific benign histopathologic finding which accounts for the presence of a lung nodule (specifically including organizing pneumonia, frank purulence, granulomatous inflammation, or other specific benign finding) AND
  * Absence of malignancy (true negative) through 1-year CT follow-up, defined as:
    * The nodule markedly regresses or resolves on follow-up imaging, OR
    * A persistent nodule has not been diagnosed as malignant, AND
    * No plans for repeat invasive diagnostic procedures through 12 months follow-up.
  Normal or absence of lung parenchyma, atypia and non-specific inflammation will be considered non-diagnostic.
Time Frame: Up to 12 months
Population: Our protocol excluded those missing primary outcome data from the primary outcome analysis. The primary outcome was adjudicated as 12 months and five patients were lost to follow-up (2 in NB group, 3 in CT-guided Biopsy group). These represent the difference in these denominators for this analysis compared to overall patient numbers. The overall patient numbers (121 an 113) were used as base denominators for all other outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 119 | 110
Participants | 94 | 81
Statistical Analysis 1: Comparison: Navigation Bronchoscopy (NB) With F-Nav vs CT-guided Biopsy; Test type: Non-Inferiority — The noninferiority margin was 10%; p = 0.003, One-sided two-sample z-test — The threshold for statistical significance was p = 0.05. The p value was not adjusted for multiple comparisons; absolute difference in percentage points = 5.4, 95% CI 2-sided [-6.5 to 17.2] — Difference in diagnostic accuracy = navigational bronchoscopy % - transthoracic biopsy %

2. Secondary Outcome: Diagnostic Yield
Description: Rate at which histopathology is obtained which explains the presence of a nodule (according to definitions set forth for the primary endpoint) and permits post-biopsy clinical decision-making without need for immediate additional diagnostic procedures.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants | 96 | 88

3. Secondary Outcome: Rate of Pneumothorax
Description: Proportion of cases complicated by pneumothorax
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants | 4 | 32

4. Secondary Outcome: Rate of Pneumothorax Requiring Chest Tube Placement
Description: Proportion of cases complicated by pneumothorax requiring chest tube placement
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants | 1 | 9

5. Secondary Outcome: Need for Hospitalization After Procedure
Description: Proportion of cases with complication necessitating hospitalization after a procedure
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants | 1 | 13

6. Secondary Outcome: Duration of Procedure
Description: Total time required to complete the procedure
Time Frame: Up to 12 months
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
minutes | 36 [28 to 47.5] | 24.5 [13 to 36]

7. Secondary Outcome: Procedural Factors Associated With Improved Yield (Type of Biopsy)
Description: Association of diagnostic yield with type of tools used to obtain biopsy: F-Nav Bronchoscopy group. This outcome measure is only applicable to the patients randomized to the navigational bronchoscopy platform.
Time Frame: Up to 12 months
Population: Total number of patients included in this analysis was 119. Two patients randomized to the bronchoscopy arm did not undergo the procedure because they had lesions that were regressing on the day of the exam. This was a pre-specified exclusion criterion in the statistical analysis plan for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Patients included are those that received the navigational bronchoscopy intervention
- Diagnostic: Patients that received a diagnostic result from the navigational bronchoscopy intervention
- Nondiagnostic: Patients that did not receive a diagnostic result from the navigational bronchoscopy intervention
Arm/Group | Overall | Diagnostic | Nondiagnostic
Number analyzed (Participants) | 119 | 94 | 25
Participants
  Transbronchial needle aspiration (TBNA) | 116 | 93 | 23
  Transbronchial biopsy (TBB) using forceps | 76 | 64 | 12
  Peripheral brushing with standard brush | 22 | 17 | 5
  Triple needle brushing | 2 | 2 | 0
  GenCut biopsy tool | 3 | 1 | 2
  Peripheral wash via navigation catheter | 31 | 22 | 9
  Any specimen cultured | 25 | 15 | 10

8. Secondary Outcome: Procedural Factors Associated With Improved Yield (Number of Biopsies)
Description: Association of diagnostic yield with count of biopsies. This outcome measure is only specific to the F-Nav bronchoscopy arm.
Time Frame: Up to 12 months
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: number of biopsies
Arm/Group | Overall | Diagnostic | Nondiagnostic
Number analyzed (Participants) | 119 | 94 | 25
number of biopsies
  TBNA needle passes | 8.0 [6.0 to 8.2] | 8.0 [6.0 to 8.0] | 8.0 [6.5 to 10.0]
  Forceps TBB pass count | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 8.0]

9. Secondary Outcome: Procedural Factors Associated With Improved Yield (Use of Radial Ultrasound)
Description: Association of diagnostic yield with use of radial ultrasound. This outcome measure is only specific to the F-Nav bronchoscopy arm.
Time Frame: Up to 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Diagnostic | Nondiagnostic
Number analyzed (Participants) | 119 | 94 | 25
Participants
  Initial Radial Endobronchial Ultrasound (REBUS) signature: Concentric | 20 | 20 | 0
  Initial REBUS signature: Eccentric | 39 | 30 | 9
  Initial REBUS signature: Could not localize | 47 | 32 | 15
  REBUS not used during procedure | 13 | 12 | 1

10. Secondary Outcome: Procedural Factors Associated With Improved Yield (Presence of a Bronchus Sign)
Description: Association of diagnostic yield with presence of a bronchus sign
Time Frame: Up to 12 months
Population: Each trial arm is being split into two groups, whether a bronchus sign was present or absent. This is sub-group analysis for each trial arm hence the different denominators. If you add the denominators for each column, it totals the overall number of participants for that trial arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants
  Presence of a bronchus sign: number analyzed (Participants) | 41 | 38
  Presence of a bronchus sign | 37 | 30
  Without a bronchus sign: number analyzed (Participants) | 80 | 75
  Without a bronchus sign | 59 | 58

11. Secondary Outcome: Procedural Factors Associated With Improved Yield (Biopsy Site)
Description: Association of diagnostic yield with biopsy site (nodule location)
Time Frame: Up to 12 months
Population: Each trial arm is being split into two groups, whether the lung nodule is in the outer-third zone or middle-third zone. This is sub-group analysis for each trial arm hence the different denominators. If you add the denominators for each column, it totals the overall number of participants for that trial arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants
  Nodule is in outer-third zone: number analyzed (Participants) | 107 | 98
  Nodule is in outer-third zone | 86 | 77
  Nodule is in middle-third zone: number analyzed (Participants) | 14 | 15
  Nodule is in middle-third zone | 10 | 11

12. Secondary Outcome: Need for Additional Nodule Biopsy
Description: Proportion of cases in which additional invasive biopsy procedures directed at the targeted nodule were subsequently performed
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants | 16 | 15

13. Secondary Outcome: Need for Additional Procedure for Staging
Description: Proportion of cases in which a subsequent procedure was performed for staging
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants | 0 | 3

14. Secondary Outcome: Radiation Exposure From Fluoroscopy-guided Bronchoscopy
Description: Count of total radiation exposure from fluoroscopy-guided bronchoscopy (units mGy*cm^2)
Time Frame: Up to 12 months
Population: The NB arm has units of mGy*cm^2.
Measure: Median (Inter-Quartile Range); unit: mGy*cm^2
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav
Number analyzed (Participants) | 121
mGy*cm^2 | 9800 [7190 to 18850]

15. Secondary Outcome: Need for F-Nav During Navigation Bronchoscopy
Description: Count of instances of need for F-Nav (digital tomosynthesis) during navigation bronchoscopy. This outcome measure pertains only for the F-Nav bronchoscopy arm.
Time Frame: Up to 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Diagnostic | Nondiagnostic
Number analyzed (Participants) | 119 | 94 | 25
Participants | 96 | 71 | 25

16. Secondary Outcome: Confident Clinical Diagnosis
Description: The proportion of biopsy procedures yielding a confident clinical diagnosis including any added yield from endobronchial ultrasound-guided mediastinal and/or hilar lymph node biopsies or microbiologic studies which yield an explanation for a nodule despite non-diagnostic biopsy specimens.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
Number analyzed (Participants) | 121 | 113
Participants | 96 | 88

17. Secondary Outcome: Radiation Exposure From CT for CT-guided Biopsy
Description: Count of total radiation exposure CT-guided transthoracic biopsy (units of mGy*cm)
Time Frame: Up to 12 months
Population: CT-guided biopsy arm has units of mGy*cm
Measure: Median (Inter-Quartile Range); unit: mGy*cm
Arm/Group | CT-guided Biopsy
Number analyzed (Participants) | 113
mGy*cm | 659 [253 to 1276]

18. Secondary Outcome: Procedural Factors Associated With Improved Yield (Type of Biopsy): CT-guided Group
Description: Association of diagnostic yield with type of tools used to obtain biopsy: CT-guided group. This outcome measure is only applicable to the patients randomized to the CT-guided procedure.
Time Frame: Up to 12 months
Population: 16 patients not included: CT performed on the day of the procedure demonstrated regressing nodules in 10 patients and the proceduralist decided to cancel in 6 patients. There were pre-specified exclusion criteria for this outcome measure.
  Two patients randomized to the bronchoscopy arm did not undergo the procedure because they had lesions that were regressing on the day of the exam. This was a pre-specified exclusion criterion in the statistical analysis plan for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Patients included are those that received the CT-guided intervention
- Diagnostic: Patients that received a diagnostic result from the CT-guided intervention
- Nondiagnostic: Patients that did not receive a diagnostic result from the CT-guided intervention
Arm/Group | Overall | Diagnostic | Nondiagnostic
Number analyzed (Participants) | 97 | 78 | 19
Participants
  Coaxial needle gauge : <19 | 6 | 4 | 2
  Coaxial needle gauge : 19 | 75 | 64 | 11
  Coaxial needle gauge : 20 | 12 | 9 | 3
  Coaxial needle gauge : Not used | 4 | 1 | 3
  FNA performed | 6 | 4 | 2
  Core biopsies performed | 89 | 78 | 11
  Core biopsy gauge: 18 or 19 | 6 | 4 | 2
  Core biopsy gauge: 20 or 21 | 83 | 74 | 9
  Any specimen cultured | 8 | 8 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Navigation Bronchoscopy (NB) With F-Nav | CT-guided Biopsy
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/113
Serious Adverse Events (participants affected / at risk) | 2/121 | 14/113
Other Adverse Events (participants affected / at risk) | 4/121 | 19/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Navigation Bronchoscopy (NB) With F-Nav (N=121) | CT-guided Biopsy (N=113)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 13
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Navigation Bronchoscopy (NB) With F-Nav (N=121) | CT-guided Biopsy (N=113)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 19
Hemorrhage requiring intervention (Blood and lymphatic system disorders) | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT04250194/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT04250194/ICF_000.pdf